CLINICAL TRIAL: NCT04530656
Title: Safety, Tolerability and Immunogenicity of a Recombinant SARS-CoV-2 Vaccine (Sf9 Cell) in Chinese Healthy Population Aged 18 Years and Older: A Phase I, Single-center, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Phase I Trial of a Recombinant SARS-CoV-2 Vaccine (Sf9 Cell)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT098
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Safety; Tolerability; Immunogenicity; SARS-CoV-2 Vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Middle-dose vaccine (18-55 years) & Two dose regimen (Experimental): Two doses of middle-dose experimental vaccine at the schedule of day 0, 28.
  Interventions: Biological: Two doses of middle-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28
- Middle-dose vaccine (> 55 years) & Two dose regimen (Experimental): Two doses of middle-dose experimental vaccine at the schedule of day 0, 28.
  Interventions: Biological: Two doses of middle-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28
- High-dose vaccine (18-55 years) & Two dose regimen (Experimental): Two doses of high-dose experimental vaccine at the schedule of day 0, 28.
  Interventions: Biological: Two doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28
- High-dose vaccine (> 55 years) & Two dose regimen (Experimental): Two doses of high-dose experimental vaccine at the schedule of day 0, 28.
  Interventions: Biological: Two doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28
- High-dose vaccine (18-55 years) & Three dose regimen (Experimental): Three doses of high-dose experimental vaccine at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 14, 28
- High-dose vaccine (> 55 years) & Three dose regimen (Experimental): Three doses of high-dose experimental vaccine at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 14, 28
- Middle-dose placebo (18-55 years) & Two dose regimen (Placebo Comparator): Two doses of middle-dose placebo at the schedule of day 0, 28.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 28（middle-dose group）
- Middle-dose placebo (> 55 years) & Two dose regimen (Placebo Comparator): Two doses of middle-dose placebo at the schedule of day 0, 28.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 28（middle-dose group）
- High-dose placebo (18-55 years) & Two dose regimen (Placebo Comparator): Two doses of high-dose placebo at the schedule of day 0, 28.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 28（high-dose group）
- High-dose placebo (> 55 years) & Two dose regimen (Placebo Comparator): Two doses of high-dose placebo at the schedule of day 0, 28.
  Interventions: Biological: Two doses of placebo at the schedule of day 0, 28（high-dose group）
- High-dose placebo (18-55 years) & Three dose regimen (Placebo Comparator): Three doses of high-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28（high-dose group）
- High-dose placebo (> 55 years) & Three dose regimen (Placebo Comparator): Three doses of high-dose placebo at the schedule of day 0, 14, 28.
  Interventions: Biological: Three doses of placebo at the schedule of day 0, 14, 28（high-dose group）

INTERVENTIONS:
Biological: Two doses of middle-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28 — Two doses of middle-dose (20µg/ 0.5ml) recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28.
  Arms: Middle-dose vaccine (18-55 years) & Two dose regimen; Middle-dose vaccine (> 55 years) & Two dose regimen
Biological: Two doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28 — Two doses of high-dose (40µg/ 1.0ml) recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 28.
  Arms: High-dose vaccine (18-55 years) & Two dose regimen; High-dose vaccine (> 55 years) & Two dose regimen
Biological: Three doses of high-dose recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 14, 28 — Three doses of high-dose (40µg/ 1.0ml) recombinant SARS-CoV-2 vaccine (Sf9 Cell) at the schedule of day 0, 14, 28
  Arms: High-dose vaccine (18-55 years) & Three dose regimen; High-dose vaccine (> 55 years) & Three dose regimen
Biological: Two doses of placebo at the schedule of day 0, 28（middle-dose group） — Two doses of placebo (0.5ml) at the schedule of day 0, 28
  Arms: Middle-dose placebo (18-55 years) & Two dose regimen; Middle-dose placebo (> 55 years) & Two dose regimen
Biological: Two doses of placebo at the schedule of day 0, 28（high-dose group） — Two doses of placebo (1.0ml) at the schedule of day 0, 28
  Arms: High-dose placebo (18-55 years) & Two dose regimen; High-dose placebo (> 55 years) & Two dose regimen
Biological: Three doses of placebo at the schedule of day 0, 14, 28（high-dose group） — Three doses of placebo (1.0ml) at the schedule of day 0, 14, 28
  Arms: High-dose placebo (18-55 years) & Three dose regimen; High-dose placebo (> 55 years) & Three dose regimen

SUMMARY:
This is a phase I, single-center, randomized, placebo-controlled, double-blind study, to evaluate safety, tolerability and immunogenicity of a recombinant SARS-CoV-2 vaccine (Sf9 cell) in Chinese healthy population aged 18 years and older. After randomization, the trial for each subject will last for approximately 13 months. Screening period is 1 week prior to randomization (Day -7 to Day -1), and each dose of either SARS-CoV-2 vaccine (Sf9 Cell) or placebo will be given intramuscularly (IM) on Day 0 and Day 28 for a two-dose regimen, or on Day 0, Day 14, and Day 28 for a three-dose regimen. Subjects who are ≥18 years old and ≤ 55 years old will be enrolled in adult group, and healthy elderly population who are >55 years old will be enrolled in elderly group. After adult group completes the follow-up 7 days after first vaccination, elderly group will be recruited.

DETAILED DESCRIPTION:
This is a phase I, single-center, randomized, placebo-controlled, double-blind study, to evaluate safety, tolerability and immunogenicity of a recombinant SARS-CoV-2 vaccine (Sf9 cell) in Chinese healthy population aged 18 years and older. Healthy adults who are ≥18 years old and ≤55 years old will be enrolled in the adult group and healthy elderly population who are >55 years old will be enrolled in the elderly group. To ensure the enrollment of healthy subjects, screening tests (hematology, biochemistry, and urinalysis) will be performed prior to the vaccination. In each age group, there are three regimen cohort: middle-dose at 0, 28 schedule, high-dose at 0, 28 schedule, and high-dose at 0,14,28 schedule. The subjects in regimen cohort will be randomized to receive vaccines or placebos at a ratio of 3:1.

The study will set up an Independent Data Monitoring Committee (IDMC) to conduct overall supervision. The IDMC is required to review the unblinded data when a significant event or risk occurs in the study that might cause the study to be suspended.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of ≥ 18 years old with body mass index (BMI) ≥ 18.5 and ≤ 30 at the Screening Visit.
* The subject can provide with informed consent and signs and dates a written informed consent form (ICF) prior to the initiation of any trial procedures.
* They must be able to understand and follow trial-related instructions.
* They must be willing and able to comply with planned visits, treatment schedule, laboratory tests and other requirements of the trial.
* Negative HIV antibody when screening.
* Axillary temperature ≤ 37.0ºC.
* Negative in nucleic acid screening of SARS-CoV-2.
* Negative in antibodies (IgG and IgM) screening of SARS-CoV-2.
* No imaging features of COVID-19 in chest CT.
* There were no significant abnormalities in blood routine, blood biochemistry, coagulation function and urine routine, or no clinical significance was determined by doctors (including white blood cell count, lymphocyte count, neutrophil count, platelet, hemoglobin, glutamic pyruvic transaminase ALT, glutamic oxaloacetic transaminase AST, total bilirubin, fasting blood glucose, creatinine, prothrombin time, partially activated prothrombin time, urine protein, urine red blood cells).
* Healthy subjects who have been examined by medical history, physical examination and clinical examination are in accordance with the immunization of this vaccine.

Exclusion Criteria:

Exclusion criteria of prime dose:

* Subjects with a medical or family history of convulsions, epilepsy, encephalopathy, and psychosis.
* Allergic to any ingredient in the study vaccine, or used to have a serious vaccine allergic reaction.
* Women who are positive for urine pregnancy test. Women who are pregnant or breastfeeding or planning to be pregnant within 6 months.
* Have acute febrile diseases or infectious diseases.
* History of SARS, SARS-CoV-2 or MERS infection.
* People with serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and can not control using drugs.
* Patients with severe chronic diseases or progressive conditions can not be smoothly controlled, such as asthma, diabetes, and thyroid diseases.
* Have congenital or acquired angioedema/neuroedema.
* Had urticaria 1 year before receiving the study vaccine.
* Asplenium or functional aspleen.
* Have thrombocytopenia or other coagulation disorders (may cause contraindications to intramuscular injection).
* Have acupuncture syncope reaction.
* Have received immunosuppressant therapy, anti-allergic therapy, cytotoxic therapy, inhaled corticosteroids in the past 6 months (excluding corticosteroid spray therapy for allergic rhinitis, and surface corticosteroid therapy for acute non-complicated dermatitis).
* Received blood products within 4 months before receiving the study vaccine.
* Received other study drugs within 1 month before receiving the study vaccine.
* Received a live attenuated vaccine within 1 month before receiving the study vaccine.
* Received a subunit or inactivated vaccine within 14 days before receiving the study vaccine.
* Are receiving anti-tuberculosis treatment.
* According to the judgment of the researchers, due to a variety of medical, psychological, social or other conditions, it is contrary to the trial scheme, or affects the subjects to sign informed consent.
* It is contrary to the trial protocol, or affects the subjects to sign informed consent due to various medical, psychological, social or other conditions, according to the investigator's judgment.

Exclusion criteria of subsequent dose:

* Have had a severe allergic reaction after the previous dose of vaccination.
* Those with serious adverse events that are causally related to the previous dose of vaccination.
* For those newly discovered or occurred after the prime vaccination that does not meet the prime-dose inclusion criteria or meets the prime-dose exclusion criteria, it is up to the investigator to determine whether to continue to participate in the study or not.
* Other exclusion reasons determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions (AR) within 7 days after each dose of the recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo. | 7 days after each dose.
  Occurrence of solicited AR in the subjects within 7 days after each dose of recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo.

SECONDARY OUTCOMES:
Occurrence of adverse events (AE) within 7 days after each dose of the recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo. | 7 days after each dose.
  Occurrence of solicited AE in the subjects within 7 days after each dose of recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo.
Occurrence of AE up to Day 28 after prime and boost vaccination. | Day 28 after prime and boost vaccination.
  Occurrence of subjects experiencing AE associated with recombinant SARS-CoV-2 vaccine (Sf9 cell) up to Day 28.
The proportion of SAEs up to Day 28 after prime and boost vaccination. | Day 28 after prime and boost vaccination.
  The proportion of subjects experiencing SAEs up to Day 28 after prime and boost vaccination.
The proportion of SAEs up to Month 12 after prime and boost vaccination. | The proportion of subjects experiencing SAEs up to Month 12 after prime and boost vaccination.
  Month 12 after prime and boost vaccination.
The proportion of abnormal markers of hematology, blood chemistry and urine analysis within 7 days before prime vaccination and at Day 3 after each dose of recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo. | 7 days before prime vaccination and Day 3 after each dose.
  The proportion of subjects experiencing abnormal markers of hematology, blood chemistry and urine analysis within 7 days before prime vaccination and at Day 3 after each dose of recombinant SARS-CoV-2 vaccine (Sf9 cell) or placebo.
GMT of anti-RBD specific antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Geometric mean titer (GMT) of anti-RBD specific antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
Four-fold increase in anti-RBD specific antibody titers, at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Four-fold increase in anti-RBD specific antibody titers, as compared to baseline, at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
GMFI of anti-RBD specific antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Geometric mean fold increase (GMFI) of anti-RBD specific antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
GMT of SARS-CoV-2 neutralizing antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody (including pseudovirus and live virus-based SARS-CoV-2 neutralizing antibody assay) at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after prime and boost vaccination.
Four-fold increase in SARS-CoV-2 neutralizing antibody titers, at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Four-fold increase in SARS-CoV-2 neutralizing antibody titers (including pseudovirus and live virus-based SARS-CoV-2 neutralizing antibody assay), as compared to baseline, at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
GMFI of SARS-CoV-2 neutralizing antibody at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after prime and boost vaccination. | Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
  Geometric mean fold increase (GMFI) of SARS-CoV-2 neutralizing antibody (including pseudovirus and live virus-based SARS-CoV-2 neutralizing antibody assay) at Day 7, Day 14, Day 28, Month 3, Month 6, and Month 12 after boost vaccination.
Seroconversion rates of IFN-γ stimulated by the overlapping peptide library of S-RBD protein at Day 14, Day 28 after boost vaccination. | Day 14, Day 28 after boost vaccination.
  Seroconversion rates of IFN-γ stimulated by the overlapping peptide library of S-RBD protein at Day 14, Day 28 after boost vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China